CLINICAL TRIAL: NCT03319940
Title: A Phase 1 Study Evaluating the Safety, Tolerability and Pharmacokinetics of Tarlatamab in Subjects With Small Cell Lung Cancer (DeLLphi-300)
Brief Title: Study Evaluating Safety, Tolerability and Pharmacokinetics (PK) of Tarlatamab in Adults With Small Cell Lung Cancer (SCLC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160323
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2017-10-05; First posted 2017-10-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Half-Life Extended (HLE) Bispecific T cell engager (BiTE®); Delta-like protein 3 (DLL3); Tarlatamab; Oncology; Immunology
MeSH Terms: conditions — Small Cell Lung Carcinoma; Bites and Stings; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, ascending, multiple doses, phase 1 study evaluating tarlatamab monotherapy, in combination with anti-PD1 therapy and with additional CRS mitigation strategies in participants with SCLC. The dose exploration phases of the study will estimate the maximum tolerated dose (MTD) or Recommended Phase 2 Dose (RP2D) of tarlatamab either as monotherapy or in combination with pembrolizumab. This will be followed by dose expansion phase to confirm RP2D and to obtain further safety and efficacy data.
Masking Description: The patient, investigator, investigative staff, medical monitor and care provider will not be masked for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Experimental): Tarlatamab monotherapy
  Interventions: Drug: Tarlatamab
- Part C (Experimental): Tarlatamab with Pembrolizumab
  Interventions: Drug: Tarlatamab; Drug: Pembrolizumab
- Part D (Experimental): Tarlatamab with additional CRS mitigation strategies
  Interventions: Drug: Tarlatamab; Drug: CRS Mitigation Strategies
- Part E (Experimental): Tarlatamab administration with 24-hour monitoring
  Interventions: Drug: Tarlatamab
- Part F (Experimental): Tarlatamab administered in outpatient infusion centers with 8-hour monitoring
  Optional wearable digital device substudy (US sites only)
  Interventions: Drug: Tarlatamab
- Part G (Experimental): Tarlatamab additional dosing schedule
  Optional wearable digital device substudy (US sites only)
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab is a Half-Life Extended (HLE) Bispecific T cell engager (BiTE®) targeting delta-like protein 3 (DLL3)
Drug: Pembrolizumab — Pembrolizumab is a potent humanized IgG4 monoclonal antibody (mAb) with high specificity of binding to the PD-1 receptor, thus inhibiting its interaction with PD-L1 and PD-L2
  Arms: Part C
Drug: CRS Mitigation Strategies — Participants will be treated with one of the CRS mitigation strategies.
  Arms: Part D

SUMMARY:
A study to assess the safety, tolerability, and PK of tarlatamab in participants with SCLC

DETAILED DESCRIPTION:
This is an open-label, ascending, multiple doses, phase 1 study evaluating tarlatamab monotherapy, in combination with anti-PD1 therapy and with additional cytokine release syndrome (CRS) mitigation strategies. Tarlatamab will be administered as a short term intravenous (IV) infusion in participants with SCLC. Tarlatamab is a Half-Life Extended (HLE) Bispecific T cell engager (BiTE®) targeting delta-like protein 3 (DLL3)

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study-specific activities/procedures
* Age greater than or equal to 18 years old at the time of signing the informed consent
* Histologically or cytologically confirmed SCLC. For parts A, C, D, E, F, and G: relapsed/refractory small cell lung cancer (R/R SCLC) who progressed or recurred following platinum-based regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Participants with treated brain metastases are eligible provided they meet defined criteria
* Adequate organ function as defined in protocol

Exclusion Criteria:

* History of other malignancy within the past 2 years prior to first dose of tarlatamab with exceptions
* Major surgery within 28 days of first dose tarlatamab
* Untreated (includes new lesions or progression in previously treated lesions) or symptomatic brain metastases and leptomeningeal disease (regardless of symptomatic or not).
* Prior anti-cancer therapy: at least 28 days must have elapsed between any prior anti-cancer therapy and first dose of tarlatamab with the following exceptions: participants who received conventional chemotherapy are eligible if at least 14 days have elapsed and if all treatment-related toxicity has been resolved to Grade less than or equal to 1; and prior palliative radiotherapy must have been completed at least 7 days before the first dose of tarlatamab
* Participants who experienced severe, life-threatening or recurrent (Grade 2 or higher) immune-mediated AEs or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immune-oncology agents
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab
* Part C only: history of solid organ transplantation or active autoimmune disease that has required systemic treatment within the past 2 years
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of investigational product administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLT) for all indications | 6 months
Number of participants with treatment-emergent adverse events (AEs) for all indications | 4 years
Number of participants with treatment-related AEs for all indications | 4 years
Number of participants with clinically significant changes in vital signs for all indications | 4 years
Number of participants with significant changes in electrocardiogram (ECG) for all indications | 4 years
Number of participants with significant changes in physical examinations for all indications | 4 years
Number of participants with significant changes in clinical laboratory tests for all indications | 4 years

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) following intravenous administration for all indications | 4 years
Minimum observed concentration (Cmin) following intravenous administration for all indications | 4 years
Area under the concentration-time curve (AUC) over the 2 week dosing interval for all indications | 4 years
Accumulation following multiple dosing for all indications | 4 years
Half-life (t1/2) following intravenous administration for all indications | 4 years
Objective Response (OR) per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 4 years
  Only for parts A, D, E, F, and G
Duration of Response (DOR) for all indications | 4 years
Time to Response (TTR) | 4 years
9-month Progression-Free Survival (PFS) for all indications | 9 months
9-month Overall Survival (OS) for all indications | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (39):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - John Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - Thoracic Oncology Clinic, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Pavillion, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Chris OBrien Lifehouse, Camperdown, New South Wales, Australia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Gustave Roussy, Villejuif, France
- Universitaetsklinikum Wuerzburg, Würzburg, Germany
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Netherlands (2):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
- Poland (2):
  - Biokinetica SA, Józefów
  - Europejskie Centrum Zdrowia Otwock Szpital imienia Fryderyka Chopina, Otwock
- Spain (5):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St Gallen, Sankt Gallen
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Christie Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Owen DH, Giffin MJ, Bailis JM, Smit MD, Carbone DP, He K. DLL3: an emerging target in small cell lung cancer. J Hematol Oncol. 2019 Jun 18;12(1):61. doi: 10.1186/s13045-019-0745-2. PMID 31215500
- [Background] Dowlati A, Hummel HD, Champiat S, Olmedo ME, Boyer M, He K, Steeghs N, Izumi H, Johnson ML, Yoshida T, Bouchaab H, Borghaei H, Felip E, Jost PJ, Gadgeel S, Chen X, Yu Y, Martinez P, Parkes A, Paz-Ares L. Sustained Clinical Benefit and Intracranial Activity of Tarlatamab in Previously Treated Small Cell Lung Cancer: DeLLphi-300 Trial Update. J Clin Oncol. 2024 Oct 10;42(29):3392-3399. doi: 10.1200/JCO.24.00553. Epub 2024 Aug 29. PMID 39208379
- [Background] Paz-Ares L, Champiat S, Lai WV, Izumi H, Govindan R, Boyer M, Hummel HD, Borghaei H, Johnson ML, Steeghs N, Blackhall F, Dowlati A, Reguart N, Yoshida T, He K, Gadgeel SM, Felip E, Zhang Y, Pati A, Minocha M, Mukherjee S, Goldrick A, Nagorsen D, Hashemi Sadraei N, Owonikoko TK. Tarlatamab, a First-in-Class DLL3-Targeted Bispecific T-Cell Engager, in Recurrent Small-Cell Lung Cancer: An Open-Label, Phase I Study. J Clin Oncol. 2023 Jun 1;41(16):2893-2903. doi: 10.1200/JCO.22.02823. Epub 2023 Jan 23. PMID 36689692
- [Background] Chiang AC, Olmedo Garcia ME, Carlisle JW, Dowlati A, Reguart N, Felip E, Jost PJ, Steeghs N, Stec R, Gadgeel SM, Loong HH, Jiang W, Hamidi A, Parkes A, Paz-Ares L. Safety of tarlatamab with 6-8-h outpatient versus 48-h inpatient monitoring during cycle 1: DeLLphi-300 phase 1 substudy. ESMO Open. 2025 Apr;10(4):104538. doi: 10.1016/j.esmoop.2025.104538. Epub 2025 Apr 4. PMID 40187110
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com